CLINICAL TRIAL: NCT03452839
Title: Continuous Infusion Versus Intermittent Administration of Meropenem in Critically Ill Patients: A Multicenter Randomized Double Blind Trial
Brief Title: Bolus Versus Continuous Infusion of Meropenem
Acronym: MERCY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Full Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MERCY/9A/OSR; 2016-002052-24 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Antibiotic Resistant Infection; Critical Illness
Keywords: meropenem; antibiotic resistance; critical illness; β-lactams; continuous antibacterial drug infusion; mortality
MeSH Terms: conditions — Critical Illness | interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous infusion (Experimental): Patient randomized to continuous infusion group, will receive a continuous infusion of meropenem according to their renal function (creatinine clearance -ClCr- estimated by Cockcroft-Gault formula and study day
  1. for ClCr > 50 ml/min: 3 g / day, prepared as follows: 10 mg/ml of meropenem in NaCl 0.9% at 12,5 ml/h.
  2. for ClCr < 50 ml/min: 2 g / day, prepared as follows: 10 mg/ml of meropenem in NaCl 0.9% at 8,3 ml/h.
  This solution will be replaced every time its duration exceeds the stability in use stated by the producer
  Interventions: Drug: Meropenem
- Bolus (Active Comparator): Patient randomized to bolus group, will receive a bolus infusion of meropenem according to their renal function (creatinine clearance -ClCr- estimated by Cockcroft-Gault formula):
  1. for Cl-Cr > 50 ml/min 1 g every 6 hours on first 24 hours, every 8 hours after
  2. for Cl-Cr < 50 ml/min 1 g every 8 hours on first 24 hours, every 12 hours after
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem — Meropenem or injection vials to be re-constituted in a solution of NaCl 0.9%.

SUMMARY:
This study arises from the need to optimize antibacterial drug usage to face increasing drug resistance among gram-negative pathogens in intensive care units. Gram-negative organisms are responsible for 70% of drug-resistant infections acquired in the intensive care unit. Meropenem is a β-lactam, carbapenem, antibacterial agent usually administered by intermittent infusion. As β-lactam efficacy is determined by the time in which the drug concentration exceeds the minimum inhibiting concentration of the target pathogen, intermittent infusion of this short half-lived drug can lead to precipitous drops in serum drug levels, an occurrence linked to emergence of resistant pathogens. The investigators hypothesize a beneficial effect of a continuous meropenem infusion on mortality and emergence of drug resistant pathogens. All patients enrolled will receive 1 g of meropenem bolus. After that, subjects will be randomized to receive a continuous infusion of study drug 3g/day or a bolus administration of the same amount of drugs. The investigators expect a reduction of mortality and emergence of extensive or pan drug resistant pathogens from 52 to 40% in the continuous infusion group.

ELIGIBILITY:
Inclusion Criteria:

Will be enrolled patients who:

* Are able to express informed consent or the latter can be given by his/her next of kin or as requested by Ethical Committee.
* Need a new antibiotic treatment, by clinical judgment, with meropenem
* Are admitted to ICU
* Have Sepsis or septic shock. Sepsis defined as having all the following 1. SIRS (Systemic Inflammatory Response Syndrome); 2. suspected or documented infection; 3. a SOFA score ≥ 2. Septic shock defined as having all the following 1.Sepsis; 2. Persisting hypotension requiring vasopressors to maintain MAP ≥65mmHg and having a serum lactate level >2 mmol/L (18mg/dL) despite adequate volume resuscitation.

Exclusion Criteria:

Will be excluded patients who:

* Are able to express informed consent and deny it
* Are already receiving study drug or other carbapenem both as a bolus or continuous infusion
* Have a known allergy or intolerance to study drug, to other carbapenem antibacterial agents or severe allergic reaction to β-lactam antibacterial agents or to anhydrous sodium carbonate (study drug excipient)
* Have a little chance of survival, as defined by a SAPS II score greater than 65
* Have concomitant acquired immunodeficiency syndrome (stage 3 according to CDC)
* Received immunosuppressant or long-term corticosteroid therapy (more than 0.5 mg/kg/day for over 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Death or Emergence of new resistant bacteria | day 28
  composite outcome:
  1. death from any cause at day 28
  2. emergence of new XDR (extended drug resistant) or PDR (pan drug resistant) bacteria at day 28

SECONDARY OUTCOMES:
Death from any cause | day 90
  Death from any cause
Antibiotic-free days | up to day 28 or death
  Proportion of days from randomization to day 28 or death in which subject didn't receive any antibiotics (excluding anti-fungal anti-viral drugs)
ICU - free days | day 28 or death
  Number of days from randomization to day 28 (or death) in which the subject is outside the ICU. For any discharge lasting less than 48h, no ICU-free day will be computed. Re-admission lasting less than 24 hours will not reduce ICU-free days. Patients that will not survive outside ICU for at least 48 hours, will have a ICU-free day of zero
Cumulative SOFA-free point | up to day 28
  SOFA score will be evaluated every day up to day 28. SOFA-free daily score is 24 (maximum SOFA) minus actual SOFA. Cumulative SOFA-free is the sum of SOFA-free daily from randomization to date 28. Patients dead before day 28 can't ameliorate their SOFA-free score. This way, the higher the cumulative SOFA-free, the higher is the amelioration of the patient and his probability of survival.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zangrillo, Prof, Principal Investigator — IRCCS San Raffaele Scientific Institute; Giacomo Monti, MD, Study Chair — IRCCS San Raffaele Scientific Institute
Locations (26):
- University Hospital Dubrava, Dubrava, Croatia
- Italy (22):
  - Città di Lecce Hospital, Lecce, Apulia
  - ASST Cremona, Cremona, Cemona
  - Policlinico Univeristario Campus Bio-Medico, Rome, Lazio
  - Ospedale San Raffaele di Milano, Milan, MI
  - A.O.U. Mater Domini, Catanzaro, Reggio Calabria
  - Azienda Ospedaliera Universitaria, Cagliari, Sardinia
  - USSL 10 Veneto, San Donà di Piave, Venezia
  - Ospedale San Lazzaro ASL CN2, Alba
  - Ospedale A. Cardarelli, Campobasso
  - P.O. Pineta Grande - Castelvolturno, Caserta
  - Azienda Ospedaliero Universitaria Careggi - Firenze, Florence
  - Azienda Universitario-Ospedaliera O.O.R.R., Foggia
  - E. O. Ospedali Galliera, Genova
  - Ospedale di Merano, Merano
  - Università degli Studi della Campania "L. Vanvitelli, Napoli
  - Azienda Ospedale - Università Padova - Ospedale "Sant'Antonio, Padua
  - AOU Pisana, Pisa
  - A.O.R San Carlo, Potenza
  - Grande Ospedale Metropolitano, Reggio Calabria
  - Humanitas Research Hospital, Rozzano
  - AO Città della Salute e della Scienza, Torino
  - Università di Udine, Udine
- Astana Medical University, Kazakhstan, Kazakhstan
- Russia (2):
  - Federal Clinical & Research Center for Reanimatology and Rehabilitation, Moscow
  - I.M. Sechenov Firts Moscow State Medical, Moscow

REFERENCES:
- [Background] Monti G, Galbiati C, Toffoletto F, Calabro MG, Colombo S, Ferrara B, Giardina G, Lembo R, Marzaroli M, Moizo E, Mucci M, Pasculli N, Plumari VP, Scandroglio AM, Tozzi M, Momesso E, Boffa N, Lobreglio R, Montrucchio G, Guarracino F, Benedetto U, Biondi-Zoccai G, D'Ascenzo F, D'Andrea N, Paternoster G, Ananiadou S, Ballestra M, De Sio A, Pota V, Cotoia A, Della Selva A, Bruni A, Iapichino G, Bradic N, Corradi F, Gemma M, Nogtev P, Petrova M, Agro FE, Cabrini L, Forfori F, Likhvantsev V, Bove T, Finco G, Landoni G, Zangrillo A; Collaborators. Continuous infusion versus intermittent administration of meropenem in critically ill patients (MERCY): A multicenter randomized double-blind trial. Rationale and design. Contemp Clin Trials. 2021 May;104:106346. doi: 10.1016/j.cct.2021.106346. Epub 2021 Mar 6. PMID 33684595
- [Result] Monti G, Bradic N, Marzaroli M, Konkayev A, Fominskiy E, Kotani Y, Likhvantsev VV, Momesso E, Nogtev P, Lobreglio R, Redkin I, Toffoletto F, Bruni A, Baiardo Redaelli M, D'Andrea N, Paternoster G, Scandroglio AM, Gallicchio F, Ballestra M, Calabro MG, Cotoia A, Perone R, Cuffaro R, Montrucchio G, Pota V, Ananiadou S, Lembo R, Musu M, Rauch S, Galbiati C, Pinelli F, Pasin L, Guarracino F, Santarpino G, Agro FE, Bove T, Corradi F, Forfori F, Longhini F, Cecconi M, Landoni G, Bellomo R, Zangrillo A; MERCY Investigators. Continuous vs Intermittent Meropenem Administration in Critically Ill Patients With Sepsis: The MERCY Randomized Clinical Trial. JAMA. 2023 Jul 11;330(2):141-151. doi: 10.1001/jama.2023.10598. PMID 37326473